CLINICAL TRIAL: NCT00422058
Title: Effect of Liraglutide on Body Weight in Obese Subjects Without Diabetes: A 20-week Randomised, Double-blind, Placebo-controlled, Six Armed Parallel Group, Multi-centre, Multinational Trial With an Open Label Orlistat Comparator Arm and With an 84-week Extension Period
Brief Title: The Effect of Liraglutide on Body Weight in Obese Subjects Without Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NN8022-1807; 2006-004481-13 (EudraCT Number); NCT00480909 (obsolete NCT alias)
Record Dates: First submitted 2007-01-12; First posted 2007-01-15 (Estimated); Results first posted 2010-10-28 (Estimated); Last update posted 2017-11-01 (Actual); Status verified 2017-09

CONDITIONS: Metabolism and Nutrition Disorder; Obesity
MeSH Terms: conditions — Nutrition Disorders; Obesity | interventions — Liraglutide; Orlistat

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Lira placebo/Lira 2.4 mg/Lira 3.0 mg (Placebo Comparator): Liraglutide placebo once daily, weeks 0-20 (double-blinded), extended to 52 weeks (sponsor was unblinded at 20 weeks). Subjects switched to receive liraglutide 2.4 mg once daily and then liraglutide 3.0 mg once daily in open-label extension period (weeks 52-104)
  Interventions: Drug: placebo
- Lira 1.2 mg/Lira 3.0 mg (Experimental): Liraglutide 1.2 mg once daily, weeks 0-20 (double-blinded), extended to 52 weeks (sponsor was unblinded at 20 weeks). Subjects switched to receive liraglutide 2.4 mg once daily and then liraglutide 3.0 mg once daily in open-label extension period (weeks 52-104)
  Interventions: Drug: liraglutide
- Lira 1.8 mg/Lira 3.0 mg (Experimental): Liraglutide 1.8 mg once daily, weeks 0-20 (double-blinded), extended to 52 weeks (sponsor was unblinded at 20 weeks). Subjects switched to receive liraglutide 2.4 mg once daily and then liraglutide 3.0 mg once daily in open-label extension period (weeks 52-104)
  Interventions: Drug: liraglutide
- Lira 2.4 mg/Lira 3.0 mg (Experimental): Liraglutide 2.4 mg once daily, weeks 0-20 (double-blinded), extended to 52 weeks (sponsor was unblinded at 20 weeks). Subjects switched to receive liraglutide 2.4 mg once daily and then liraglutide 3.0 mg once daily in open-label extension period (weeks 52-104)
  Interventions: Drug: liraglutide
- Liraglutide 3.0 mg (Experimental): Liraglutide 3.0 mg once daily, weeks 0-20 (double-blinded), extended to 52 weeks (sponsor was unblinded at 20 weeks). Subjects switched to receive liraglutide 2.4 mg once daily and then liraglutide 3.0 mg once daily in open-label extension period (weeks 52-104)
  Interventions: Drug: liraglutide; Drug: placebo
- Orlistat (Active Comparator): Orlistat capsules 3 times daily (3 x 120 mg) in connection with each main meal, weeks 0-20 (open-label) continued to receive Orlistat capsules 3 times daily (3 x 120 mg) in connection with each main meal in open-label extension period (weeks 20-104)
  Interventions: Drug: orlistat

INTERVENTIONS:
Drug: liraglutide — Injected s.c. (under the skin) once daily
  Arms: Lira 1.2 mg/Lira 3.0 mg; Lira 1.8 mg/Lira 3.0 mg; Lira 2.4 mg/Lira 3.0 mg; Liraglutide 3.0 mg
Drug: orlistat — 120 mg capsule. Administered thrice daily
  Arms: Orlistat
Drug: placebo — Injected s.c. (under the skin) once daily
  Arms: Lira placebo/Lira 2.4 mg/Lira 3.0 mg; Liraglutide 3.0 mg

SUMMARY:
This trial is conducted in Europe. The purpose of the 20-week trial is to investigate the efficacy of liraglutide to induce body weight loss and the purpose of the extension is to evaluate the long term safety and tolerability of liraglutide.

Trial has the following trial periods: A 20-week randomised, double-blind, placebo-controlled, six-armed parallel-group, multi-centre, multinational trial with an open label orlistat comparator arm followed by an 84 week extension period.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) greater than or equal to 30.0 or lesser than or equal to 40.0 kg/m2
* Stable body weight (less than 5% selfreported change within the last 3 months)

Exclusion Criteria:

* Obesity induced by drug treatment
* Use of approved drugs for weight lowering intervention (e.g. orlistat, sibutramin, rimonabant) within the last 3 months prior to entering trial
* Type 1 or type 2 diabetes

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 564 (Actual)
Dates: Start 2007-01-10 (Actual); Primary Completion 2007-09-13 (Actual); Study Completion 2009-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (17):
- Novo Nordisk Investigational Site, Edegem, Belgium
- Novo Nordisk Investigational Site, Prague, Czechia
- Denmark (3):
  - Novo Nordisk Investigational Site, Århus C
  - Novo Nordisk Investigational Site, Frederiksberg C
  - Novo Nordisk Investigational Site, Hvidovre
- Finland (3):
  - Novo Nordisk Investigational Site, Helsinki
  - Novo Nordisk Investigational Site, Kuopio
  - Novo Nordisk Investigational Site, Oulu
- Novo Nordisk Investigational Site, Almere Stad, Netherlands
- Spain (3):
  - Novo Nordisk Investigational Site, Barcelona
  - Novo Nordisk Investigational Site, Madrid
  - Novo Nordisk Investigational Site, Pamplona
- Sweden (2):
  - Novo Nordisk Investigational Site, Malmo
  - Novo Nordisk Investigational Site, Stockholm
- United Kingdom (3):
  - Novo Nordisk Investigational Site, Glasgow
  - Novo Nordisk Investigational Site, Luton
  - Novo Nordisk Investigational Site, Norwich

REFERENCES:
- [Result] Astrup A, Carraro R, Finer N, Harper A, Kunesova M, Lean ME, Niskanen L, Rasmussen MF, Rissanen A, Rossner S, Savolainen MJ, Van Gaal L; NN8022-1807 Investigators. Safety, tolerability and sustained weight loss over 2 years with the once-daily human GLP-1 analog, liraglutide. Int J Obes (Lond). 2012 Jun;36(6):843-54. doi: 10.1038/ijo.2011.158. Epub 2011 Aug 16. PMID 21844879
- [Result] Astrup A, Rossner S, Van Gaal L, Rissanen A, Niskanen L, Al Hakim M, Madsen J, Rasmussen MF, Lean ME; NN8022-1807 Study Group. Effects of liraglutide in the treatment of obesity: a randomised, double-blind, placebo-controlled study. Lancet. 2009 Nov 7;374(9701):1606-16. doi: 10.1016/S0140-6736(09)61375-1. Epub 2009 Oct 23. PMID 19853906
- [Result] Lean ME, Carraro R, Finer N, Hartvig H, Lindegaard ML, Rossner S, Van Gaal L, Astrup A; NN8022-1807 Investigators. Tolerability of nausea and vomiting and associations with weight loss in a randomized trial of liraglutide in obese, non-diabetic adults. Int J Obes (Lond). 2014 May;38(5):689-97. doi: 10.1038/ijo.2013.149. Epub 2013 Aug 14. PMID 23942319
- [Result] Steinberg WM, Rosenstock J, Wadden TA, Donsmark M, Jensen CB, DeVries JH. Impact of Liraglutide on Amylase, Lipase, and Acute Pancreatitis in Participants With Overweight/Obesity and Normoglycemia, Prediabetes, or Type 2 Diabetes: Secondary Analyses of Pooled Data From the SCALE Clinical Development Program. Diabetes Care. 2017 Jul;40(7):839-848. doi: 10.2337/dc16-2684. Epub 2017 May 4. PMID 28473337
- [Result] O'Neil PM, Aroda VR, Astrup A, Kushner R, Lau DCW, Wadden TA, Brett J, Cancino AP, Wilding JPH; Satiety and Clinical Adiposity - Liraglutide Evidence in individuals with and without diabetes (SCALE) study groups. Neuropsychiatric safety with liraglutide 3.0 mg for weight management: Results from randomized controlled phase 2 and 3a trials. Diabetes Obes Metab. 2017 Nov;19(11):1529-1536. doi: 10.1111/dom.12963. Epub 2017 Jul 21. PMID 28386912
- [Result] Davies MJ, Aronne LJ, Caterson ID, Thomsen AB, Jacobsen PB, Marso SP; Satiety and Clinical Adiposity - Liraglutide Evidence in individuals with and without diabetes (SCALE) study groups. Liraglutide and cardiovascular outcomes in adults with overweight or obesity: A post hoc analysis from SCALE randomized controlled trials. Diabetes Obes Metab. 2018 Mar;20(3):734-739. doi: 10.1111/dom.13125. Epub 2017 Nov 1. PMID 28950422
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 19 sites in 8 countries: Denmark (3), Sweden (2), Finland (3), UK (3), Netherlands (1), Belgium (1), Spain (4) and Czech Republic (2)
Pre-assignment Details: Between screening and randomisation, eligible subjects were included in a 2-week single-blind run-in period in which all subjects were placed on a hypocaloric diet. The dose of liraglutide and placebo was increased during the first 4 weeks after randomisation until maintenance dose was reached. Orlistat dose was fixed from randomisation.
Period: Double-Blind, Week 0-20
Arm/Group | Lira Placebo/Lira 2.4 mg/Lira 3.0 mg | Lira 1.2 mg/Lira 3.0 mg | Lira 1.8 mg/Lira 3.0 mg | Lira 2.4 mg/Lira 3.0 mg | Liraglutide 3.0 mg | Orlistat
Started | 98 | 95 | 90 | 93 | 93 | 95
Completed | 79 | 85 | 74 | 73 | 82 | 79
Not Completed | 19 | 10 | 16 | 20 | 11 | 16
Not completed — Adverse Event | 3 | 4 | 5 | 9 | 5 | 3
Not completed — Protocol Violation | 3 | 2 | 2 | 3 | 2 | 2
Not completed — Lack of Efficacy | 2 | 1 | 1 | 0 | 0 | 1
Not completed — Other | 11 | 3 | 8 | 8 | 4 | 10
Period: Open-Label Extension, Week 20-104
Arm/Group | Lira Placebo/Lira 2.4 mg/Lira 3.0 mg | Lira 1.2 mg/Lira 3.0 mg | Lira 1.8 mg/Lira 3.0 mg | Lira 2.4 mg/Lira 3.0 mg | Liraglutide 3.0 mg | Orlistat
Started | 79 | 85 | 74 | 73 | 82 | 79
Enrolled in Extension | 67 | 68 | 59 | 65 | 72 | 67
Completed | 47 | 46 | 38 | 45 | 47 | 45
Not Completed | 32 | 39 | 36 | 28 | 35 | 34
Not completed — Not giving consent for extension | 12 | 17 | 15 | 8 | 10 | 12
Not completed — Adverse Event | 3 | 4 | 7 | 4 | 4 | 0
Not completed — Protocol Violation | 1 | 2 | 3 | 1 | 5 | 3
Not completed — Lack of Efficacy | 3 | 2 | 5 | 2 | 0 | 1
Not completed — Other | 13 | 14 | 6 | 13 | 16 | 18

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lira Placebo/Lira 2.4 mg/Lira 3.0 mg | Lira 1.2 mg/Lira 3.0 mg | Lira 1.8 mg/Lira 3.0 mg | Lira 2.4 mg/Lira 3.0 mg | Liraglutide 3.0 mg | Orlistat | Total
Number analyzed (Participants) | 98 | 95 | 90 | 93 | 93 | 95 | 564
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.86 (10.28) | 47.18 (9.72) | 45.53 (10.9) | 45.01 (11.09) | 45.91 (10.71) | 45.94 (9.11) | 45.91 (10.29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 74 | 73 | 68 | 71 | 70 | 73 | 429
  Male | 24 | 22 | 22 | 22 | 23 | 22 | 135
Race/Ethnicity, Customized [Number; unit: participants]
  White | 97 | 94 | 88 | 91 | 92 | 93 | 555
  American Indian/Alaska Native | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Black/African American | 1 | 0 | 2 | 1 | 1 | 1 | 6
  Other | 0 | 1 | 0 | 1 | 0 | 0 | 2
BMI [Mean (Standard Deviation); unit: kg/m^2] — BMI = Body Mass Index
  kg/m^2 | 34.9 (2.8) | 34.8 (2.6) | 35.0 (2.6) | 35.0 (2.8) | 34.8 (2.8) | 34.1 (2.6) | 34.8 (2.7)
Weight [Mean (Standard Deviation); unit: kg] | 97.3 (12.3) | 96.2 (13.5) | 98.0 (12.5) | 98.4 (13.0) | 97.6 (13.7) | 96.0 (11.7) | 97.2 (12.8)
Waist circumference [Mean (Standard Deviation); unit: cm] | 108.3 (10.0) | 108.8 (10.4) | 108.2 (9.5) | 110.2 (10.7) | 108.9 (8.3) | 107.6 (9.7) | 108.7 (9.8)
HbA1c [Mean (Standard Deviation); unit: percentage (%) of total haemoglobin] — HbA1c = glycosylated haemoglobin A1c
  percentage (%) of total haemoglobin | 5.60 (0.38) | 5.58 (0.33) | 5.60 (0.40) | 5.54 (0.33) | 5.57 (0.40) | 5.55 (0.32) | 5.60 (0.4)
Blood pressure [Mean (Standard Deviation); unit: mmHg]
  Systolic | 123.6 (11.1) | 127.0 (13.1) | 123.4 (13.0) | 126.2 (13.9) | 124.3 (11.3) | 122.7 (13.5) | 124.5 (12.7)
  Diastolic | 76.8 (8.5) | 79.7 (9.1) | 77.9 (7.9) | 78.6 (8.2) | 77.8 (8.3) | 76.9 (7.9) | 77.9 (8.4)

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Body Weight at Week 20
Description: Calculated as mean body weight at week 20 - baseline
Time Frame: Week 0, week 20
Population: ITT (intention to treat) analysis set using LOCF (last observation carried forward) is all randomised and exposed subjects from the double-blind period, who have been exposed to at least one dose of trial product.
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Lira Placebo/Lira 2.4 mg/Lira 3.0 mg | Lira 1.2 mg/Lira 3.0 mg | Lira 1.8 mg/Lira 3.0 mg | Lira 2.4 mg/Lira 3.0 mg | Liraglutide 3.0 mg | Orlistat
Number analyzed (Participants) | 98 | 94 | 90 | 92 | 92 | 95
kg
  Baseline | 97.3 (12.3) | 96.4 (13.4) | 98.0 (12.5) | 98.4 (13.1) | 97.5 (13.8) | 96.0 (11.7)
  Change at Week 20 | -3.0 (3.3) | -5.1 (3.5) | -5.9 (5.0) | -6.6 (4.6) | -7.6 (4.6) | -4.4 (4.1)

2. Secondary Outcome: Mean Change From Baseline in Body Weight at Week 104
Description: Calculated as mean body weight at week 104 - baseline
Time Frame: Week 0, week 104
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Lira Placebo/Lira 2.4 mg/Lira 3.0 mg | Lira 1.2 mg/Lira 3.0 mg | Lira 1.8 mg/Lira 3.0 mg | Lira 2.4 mg/Lira 3.0 mg | Liraglutide 3.0 mg | Orlistat
Number analyzed (Participants) | 98 | 94 | 90 | 92 | 92 | 95
kg
  Baseline | 97.3 (12.3) | 96.4 (13.4) | 98.0 (12.5) | 98.4 (13.1) | 97.5 (13.8) | 96.0 (11.7)
  Change at Week 104 | -5.4 (5.9) | -4.9 (5.8) | -5.6 (6.5) | -6.4 (7.2) | -8.2 (7.1) | -3.8 (6.4)

3. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose at Week 20
Description: Calculated as mean fasting plasma glucose at week 20 - baseline
Time Frame: Week 0, week 20
Population: ITT (intention to treat) analysis set using (LOCF) last observation carried forward is all randomised and exposed subjects from the double-blind period, who have been exposed to at least one dose of trial product
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Lira Placebo/Lira 2.4 mg/Lira 3.0 mg | Lira 1.2 mg/Lira 3.0 mg | Lira 1.8 mg/Lira 3.0 mg | Lira 2.4 mg/Lira 3.0 mg | Liraglutide 3.0 mg | Orlistat
Number analyzed (Participants) | 92 | 88 | 84 | 89 | 86 | 89
mmol/L
  Baseline | 5.42 (0.81) | 5.30 (0.61) | 5.29 (0.56) | 5.27 (0.57) | 5.36 (0.61) | 5.3 (0.51)
  Change at Week 20 | -0.09 (0.54) | -0.39 (0.45) | -0.44 (0.63) | -0.38 (0.48) | -0.44 (0.44) | -0.10 (0.41)

4. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose at Week 104
Description: Calculated as mean fasting plasma glucose at week 104 - baseline
Time Frame: Week 0, week 104
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Lira Placebo/Lira 2.4 mg/Lira 3.0 mg | Lira 1.2 mg/Lira 3.0 mg | Lira 1.8 mg/Lira 3.0 mg | Lira 2.4 mg/Lira 3.0 mg | Liraglutide 3.0 mg | Orlistat
Number analyzed (Participants) | 92 | 88 | 84 | 89 | 86 | 89
mmol/L
  Baseline | 5.42 (0.81) | 5.30 (0.61) | 5.29 (0.56) | 5.27 (0.57) | 5.36 (0.61) | 5.30 (0.51)
  Change at Week 104 | -0.22 (0.61) | -0.09 (0.53) | -0.09 (0.64) | -0.20 (0.50) | -0.23 (0.50) | 0.02 (0.48)

5. Secondary Outcome: Change From Baseline in Fasting Insulin at Week 20
Description: Calculated as mean fasting insulin at week 20 - baseline
Time Frame: Week 0, week 20
Population: ITT (intention to treat) analysis set, only subjects with a valid assessment (LOCF, last observation carried forward not applied).
Measure: Mean (Standard Deviation); unit: pmol/L
Arm/Group | Lira Placebo/Lira 2.4 mg/Lira 3.0 mg | Lira 1.2 mg/Lira 3.0 mg | Lira 1.8 mg/Lira 3.0 mg | Lira 2.4 mg/Lira 3.0 mg | Liraglutide 3.0 mg | Orlistat
Number analyzed (Participants) | 77 | 84 | 73 | 73 | 81 | 79
pmol/L
  Baseline | 99.5 (129.2) | 82.9 (43.0) | 85.7 (49.5) | 88.7 (43.3) | 89.1 (51.9) | 85.5 (48.3)
  Change at Week 20 | -15.0 (34.0) | 8.7 (105.3) | -0.7 (48.2) | -3.9 (53.2) | -12.3 (43.3) | -16.7 (60.6)

6. Secondary Outcome: Change From Baseline in Fasting Insulin at Week 104
Description: Calculated as mean fasting insulin at week 104 - baseline
Time Frame: Week 0, week 104
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: pmol/L
Arm/Group | Lira Placebo/Lira 2.4 mg/Lira 3.0 mg | Lira 1.2 mg/Lira 3.0 mg | Lira 1.8 mg/Lira 3.0 mg | Lira 2.4 mg/Lira 3.0 mg | Liraglutide 3.0 mg | Orlistat
Number analyzed (Participants) | 44 | 42 | 33 | 42 | 44 | 39
pmol/L
  Baseline | 99.5 (129.2) | 82.9 (43.0) | 85.7 (49.5) | 88.7 (43.3) | 89.1 (51.9) | 85.5 (48.3)
  Change at Week 104 | 0.7 (53.6) | -13.5 (39.7) | 18.6 (102.6) | -2.1 (47.3) | -19.6 (44.3) | -15.3 (39.8)

7. Secondary Outcome: Change From Baseline in HbA1c (Glycosylated Haemoglobin A1c) at Week 20
Description: Calculated as mean HbA1c (glycosylated haemoglobin A1c) at week 20 - baseline
Time Frame: Week 0, week 20
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: percentage (%) of total haemoglobin
Arm/Group | Lira Placebo/Lira 2.4 mg/Lira 3.0 mg | Lira 1.2 mg/Lira 3.0 mg | Lira 1.8 mg/Lira 3.0 mg | Lira 2.4 mg/Lira 3.0 mg | Liraglutide 3.0 mg | Orlistat
Number analyzed (Participants) | 73 | 84 | 70 | 70 | 79 | 78
percentage (%) of total haemoglobin
  Baseline | 5.60 (0.38) | 5.58 (0.33) | 5.60 (0.40) | 5.54 (0.34) | 5.57 (0.40) | 5.55 (0.32)
  Change at Week 20 | 0.01 (0.22) | -0.14 (0.21) | -0.21 (0.25) | -0.22 (0.25) | -0.24 (0.29) | 0.00 (0.21)

8. Secondary Outcome: Change From Baseline in HbA1c (Glycosylated Haemoglobin A1c) at Week 104
Description: Calculated as mean HbA1c (glycosylated haemoglobin A1c) at week 104 - baseline
Time Frame: Week 0, week 104
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: percentage (%) of total haemoglobin
Arm/Group | Lira Placebo/Lira 2.4 mg/Lira 3.0 mg | Lira 1.2 mg/Lira 3.0 mg | Lira 1.8 mg/Lira 3.0 mg | Lira 2.4 mg/Lira 3.0 mg | Liraglutide 3.0 mg | Orlistat
Number analyzed (Participants) | 46 | 45 | 36 | 45 | 47 | 45
percentage (%) of total haemoglobin
  Baseline | 5.60 (0.38) | 5.58 (0.33) | 5.60 (0.40) | 5.54 (0.34) | 5.57 (0.40) | 5.55 (0.32)
  Change at Week 104 | -0.32 (0.32) | -0.25 (0.26) | -0.30 (0.22) | -0.25 (0.30) | -0.35 (0.32) | -0.18 (0.37)

9. Secondary Outcome: Change From Baseline in hsCRP (Highly Sensitive C-reactive Protein) at Week 20
Description: Calculated as mean hsCRP (highly sensitive C-reactive protein) at week 20-baseline. High hsCRP level is associated with greater cardiovascular risk
Time Frame: Week 0, week 20
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Lira Placebo/Lira 2.4 mg/Lira 3.0 mg | Lira 1.2 mg/Lira 3.0 mg | Lira 1.8 mg/Lira 3.0 mg | Lira 2.4 mg/Lira 3.0 mg | Liraglutide 3.0 mg | Orlistat
Number analyzed (Participants) | 75 | 83 | 74 | 72 | 79 | 79
mg/L
  Baseline | 3.6 (4.2) | 5.1 (6.1) | 4.4 (4.5) | 4.0 (4.2) | 3.8 (7.4) | 4.6 (4.5)
  Change at Week 20 | 0.8 (4.0) | 0.1 (8.1) | -0.8 (2.9) | 0.5 (4.7) | -1.1 (7.2) | -0.3 (4.2)

10. Secondary Outcome: Change From Baseline in hsCRP (Highly Sensitive C-reactive Protein) at Week 104
Description: Calculated as mean hsCRP (highly sensitive C-reactive protein) at week 104- baseline. High hsCRP level is associated with greater cardiovascular risk
Time Frame: Week 0, week 104
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Lira Placebo/Lira 2.4 mg/Lira 3.0 mg | Lira 1.2 mg/Lira 3.0 mg | Lira 1.8 mg/Lira 3.0 mg | Lira 2.4 mg/Lira 3.0 mg | Liraglutide 3.0 mg | Orlistat
Number analyzed (Participants) | 46 | 45 | 38 | 45 | 45 | 45
mg/L
  Baseline | 3.6 (4.2) | 5.1 (6.1) | 4.4 (4.5) | 4.0 (4.2) | 3.8 (7.4) | 4.6 (4.5)
  Change at Week 104 | -0.5 (2.6) | -1.6 (6.0) | -0.6 (8.6) | -0.9 (3.2) | -2.1 (9.3) | 2.4 (19.4)

11. Secondary Outcome: Change From Baseline in PAI-1 (Plasminogen Activator Inhibitor 1) at Week 20
Description: Calculated as mean PAI-1 (plasminogen activator inhibitor 1) at week 20-baseline. High PAI-1 is associated with greater cardiovascular risk
Time Frame: Week 0, week 20
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: U/mL
Arm/Group | Lira Placebo/Lira 2.4 mg/Lira 3.0 mg | Lira 1.2 mg/Lira 3.0 mg | Lira 1.8 mg/Lira 3.0 mg | Lira 2.4 mg/Lira 3.0 mg | Liraglutide 3.0 mg | Orlistat
Number analyzed (Participants) | 68 | 69 | 61 | 60 | 72 | 65
U/mL
  Baseline | 21.6 (9.3) | 19.5 (9.9) | 19.7 (9.8) | 17.6 (8.7) | 19.0 (9.1) | 17.4 (8.2)
  Change at Week 20 | -3.0 (8.0) | -2.0 (7.8) | -3.5 (9.5) | -2.3 (9.5) | -4.5 (8.5) | -1.2 (8.8)

12. Secondary Outcome: Change From Baseline in PAI-1 (Plasminogen Activator Inhibitor 1) at Week 104
Description: Calculated as mean PAI-1 (plasminogen activator inhibitor 1) at week 104-baseline. High PAI-1 is associated with greater cardiovascular risk
Time Frame: Week 0, week 104
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: U/mL
Arm/Group | Lira Placebo/Lira 2.4 mg/Lira 3.0 mg | Lira 1.2 mg/Lira 3.0 mg | Lira 1.8 mg/Lira 3.0 mg | Lira 2.4 mg/Lira 3.0 mg | Liraglutide 3.0 mg | Orlistat
Number analyzed (Participants) | 39 | 36 | 29 | 37 | 39 | 41
U/mL
  Baseline | 21.6 (9.3) | 19.5 (9.9) | 19.7 (9.8) | 17.6 (8.7) | 19.0 (9.1) | 17.4 (8.2)
  Change at Week 104 | -1.4 (7.0) | -0.3 (9.1) | -0.8 (9.8) | 0.3 (9.9) | 0.4 (10.9) | 2.9 (7.4)

13. Secondary Outcome: Change From Baseline in Fibrinogen at Week 20
Description: Calculated as mean fibrinogen at week 20 - baseline. High fibrinogen is associated with greater cardiovascular risk
Time Frame: Week 0, week 20
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Lira Placebo/Lira 2.4 mg/Lira 3.0 mg | Lira 1.2 mg/Lira 3.0 mg | Lira 1.8 mg/Lira 3.0 mg | Lira 2.4 mg/Lira 3.0 mg | Liraglutide 3.0 mg | Orlistat
Number analyzed (Participants) | 68 | 71 | 62 | 61 | 73 | 67
g/L
  Baseline | 3.60 (0.67) | 3.67 (0.76) | 3.75 (0.72) | 3.64 (0.72) | 3.61 (0.68) | 3.68 (0.82)
  Change at Week 20 | -0.06 (0.58) | 0.01 (0.50) | 0.02 (0.61) | 0.10 (0.69) | 0.05 (0.55) | -0.12 (0.75)

14. Secondary Outcome: Change From Baseline in Fibrinogen at Week 104
Description: Calculated as mean fibrinogen at week 104 - baseline. High fibrinogen is associated with greater cardiovascular risk
Time Frame: Week 0, week 104
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Lira Placebo/Lira 2.4 mg/Lira 3.0 mg | Lira 1.2 mg/Lira 3.0 mg | Lira 1.8 mg/Lira 3.0 mg | Lira 2.4 mg/Lira 3.0 mg | Liraglutide 3.0 mg | Orlistat
Number analyzed (Participants) | 39 | 38 | 29 | 36 | 39 | 41
g/L
  Baseline | 3.60 (0.67) | 3.67 (0.76) | 3.75 (0.72) | 3.64 (0.72) | 3.61 (0.68) | 3.68 (0.82)
  Change at Week 104 | -0.10 (0.74) | -0.14 (0.73) | -0.15 (0.98) | -0.24 (0.74) | -0.22 (0.82) | -0.39 (1.24)

15. Secondary Outcome: Change From Baseline in Adiponectin at Week 20
Description: Calculated as mean adiponectin at week 20-baseline. A low adiponectin level is associated with greater cardiovascular risk
Time Frame: Week 0, week 20
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Lira Placebo/Lira 2.4 mg/Lira 3.0 mg | Lira 1.2 mg/Lira 3.0 mg | Lira 1.8 mg/Lira 3.0 mg | Lira 2.4 mg/Lira 3.0 mg | Liraglutide 3.0 mg | Orlistat
Number analyzed (Participants) | 77 | 82 | 72 | 70 | 79 | 77
mcg/mL
  Baseline | 5.1 (3.8) | 5.8 (3.8) | 6.7 (4.6) | 6.2 (4.6) | 6.1 (4.0) | 5.4 (4.7)
  Change at Week 20 | 2.3 (5.0) | 1.2 (5.0) | 1.7 (6.9) | 1.6 (5.7) | 2.3 (4.6) | 1.7 (4.4)

16. Secondary Outcome: Change From Baseline in Adiponectin at Week 104
Description: Calculated as mean adiponectin at week 104-baseline. A low adiponectin level is associated with greater cardiovascular risk
Time Frame: Week 0, week 104
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Lira Placebo/Lira 2.4 mg/Lira 3.0 mg | Lira 1.2 mg/Lira 3.0 mg | Lira 1.8 mg/Lira 3.0 mg | Lira 2.4 mg/Lira 3.0 mg | Liraglutide 3.0 mg | Orlistat
Number analyzed (Participants) | 39 | 36 | 27 | 39 | 35 | 39
mcg/mL
  Baseline | 5.1 (3.8) | 5.8 (3.8) | 6.7 (4.6) | 6.2 (4.6) | 6.1 (4.0) | 5.4 (4.7)
  Change at Week 104 | 3.5 (4.4) | 3.3 (3.8) | 1.3 (3.9) | 3.4 (5.4) | 3.2 (4.1) | 3.1 (4.2)

17. Secondary Outcome: Change From Baseline in Waist Circumference at Week 20
Description: Calculated as mean waist circumference at week 20-baseline.
Time Frame: Week 0, week 20
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Lira Placebo/Lira 2.4 mg/Lira 3.0 mg | Lira 1.2 mg/Lira 3.0 mg | Lira 1.8 mg/Lira 3.0 mg | Lira 2.4 mg/Lira 3.0 mg | Liraglutide 3.0 mg | Orlistat
Number analyzed (Participants) | 90 | 93 | 83 | 85 | 85 | 87
cm
  Baseline | 108.3 (10.0) | 109.0 (10.3) | 108.2 (9.5) | 110.4 (10.6) | 108.7 (8.3) | 107.6 (9.7)
  Change at Week 20 | -4.2 (4.7) | -5.8 (6.1) | -5.9 (5.3) | -7.2 (5.8) | -7.9 (5.5) | -6.0 (5.4)

18. Secondary Outcome: Change From Baseline in Waist Circumference at Week 104
Description: Calculated as mean waist circumference at week 104-baseline.
Time Frame: Week 0, week 104
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Lira Placebo/Lira 2.4 mg/Lira 3.0 mg | Lira 1.2 mg/Lira 3.0 mg | Lira 1.8 mg/Lira 3.0 mg | Lira 2.4 mg/Lira 3.0 mg | Liraglutide 3.0 mg | Orlistat
Number analyzed (Participants) | 47 | 46 | 38 | 45 | 47 | 45
cm
  Baseline | 108.3 (10.0) | 109.0 (10.3) | 108.2 (9.5) | 110.4 (10.6) | 108.7 (8.3) | 107.6 (9.7)
  Change at Week 104 | -10.0 (7.2) | -8.6 (7.5) | -9.0 (8.7) | -10.4 (7.8) | -9.8 (7.5) | -9.5 (7.3)

19. Secondary Outcome: Change From Baseline in Blood Pressure at Week 20
Description: Calculated as mean blood pressure at week 20-baseline.
Time Frame: Week 0, week 20
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Lira Placebo/Lira 2.4 mg/Lira 3.0 mg | Lira 1.2 mg/Lira 3.0 mg | Lira 1.8 mg/Lira 3.0 mg | Lira 2.4 mg/Lira 3.0 mg | Liraglutide 3.0 mg | Orlistat
Number analyzed (Participants) | 94 | 88 | 85 | 89 | 89 | 90
mmHg
  Baseline (Systolic ) | 123.6 (11.1) | 127.2 (13.1) | 123.4 (13.0) | 126.3 (13.9) | 124.3 (11.3) | 122.7 (13.5)
  Change at Week 20 (Systolic) | -3.2 (13.3) | -6.1 (11.1) | -4.8 (12.7) | -9.1 (12.3) | -6.4 (10.0) | -4.3 (10.9)
  Baseline (Diastolic) | 76.78 (8.50) | 79.71 (9.12) | 77.91 (7.92) | 78.53 (8.23) | 77.84 (8.38) | 76.94 (7.94)
  Change at Week 20 (Diastolic) | -0.32 (7.52) | -1.53 (9.15) | -1.61 (8.04) | -1.39 (7.79) | -2.37 (7.71) | -1.96 (7.82)

20. Secondary Outcome: Change From Baseline in Blood Pressure at Week 104
Description: Calculated as mean blood pressure at week 104-baseline.
Time Frame: Week 0, week 104
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Lira Placebo/Lira 2.4 mg/Lira 3.0 mg | Lira 1.2 mg/Lira 3.0 mg | Lira 1.8 mg/Lira 3.0 mg | Lira 2.4 mg/Lira 3.0 mg | Liraglutide 3.0 mg | Orlistat
Number analyzed (Participants) | 94 | 88 | 85 | 89 | 89 | 90
mmHg
  Baseline (Systolic ) | 123.6 (11.1) | 127.2 (13.1) | 123.4 (13.0) | 126.3 (13.9) | 124.3 (11.3) | 122.7 (13.5)
  Change at Week 104 (Systolic) | -2.0 (13.8) | -4.0 (13.4) | -3.8 (16.0) | -6.5 (12.6) | -5.6 (11.7) | -2.0 (11.7)
  Baseline (Diastolic) | 76.78 (8.50) | 79.71 (9.12) | 77.91 (7.92) | 78.53 (8.23) | 77.84 (8.38) | 76.94 (7.94)
  Change at Week 104 (Diastolic) | 1.64 (8.47) | -0.98 (9.81) | -1.00 (9.37) | -1.99 (9.61) | -1.92 (9.41) | -1.11 (8.36)

ADVERSE EVENTS:
Time Frame: The adverse events were collected over 104 weeks.
Description: Safety analysis set consists of all subjects exposed to trial product(s).
Arm/Group | Lira Placebo/Lira 2.4 mg/Lira 3.0 mg | Lira 1.2 mg/Lira 3.0 mg | Lira 1.8 mg/Lira 3.0 mg | Lira 2.4 mg/Lira 3.0 mg | Liraglutide 3.0 mg | Orlistat
Serious Adverse Events (participants affected / at risk) | 6/98 | 9/95 | 10/90 | 7/93 | 10/93 | 6/95
Other Adverse Events (participants affected / at risk) | 90/98 | 90/95 | 86/90 | 89/93 | 90/93 | 89/95
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lira Placebo/Lira 2.4 mg/Lira 3.0 mg (N=98) | Lira 1.2 mg/Lira 3.0 mg (N=95) | Lira 1.8 mg/Lira 3.0 mg (N=90) | Lira 2.4 mg/Lira 3.0 mg (N=93) | Liraglutide 3.0 mg (N=93) | Orlistat (N=95)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Colitis ulcerative (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hernial eventration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Abscess limb (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Post procedural infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anaesthetic complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Foreign body trauma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Multiple injuries (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ligament calcification (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Stress urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bundle branch block left (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thyroglossal cyst (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vestibular neuronitis (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Retinal detachment (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ovarian cyst ruptured (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lira Placebo/Lira 2.4 mg/Lira 3.0 mg (N=98) | Lira 1.2 mg/Lira 3.0 mg (N=95) | Lira 1.8 mg/Lira 3.0 mg (N=90) | Lira 2.4 mg/Lira 3.0 mg (N=93) | Liraglutide 3.0 mg (N=93) | Orlistat (N=95)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 6 (6) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (5)
Abdominal distension (Gastrointestinal disorders) | 5 (5) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 6 (6) | 0 (0) | 6 (6) | 0 (0) | 0 (0) | 7 (10)
Abdominal pain upper (Gastrointestinal disorders) | 5 (6) | 6 (9) | 0 (0) | 5 (6) | 7 (9) | 8 (10)
Constipation (Gastrointestinal disorders) | 15 (19) | 20 (24) | 12 (14) | 22 (29) | 19 (23) | 7 (9)
Diarrhoea (Gastrointestinal disorders) | 20 (27) | 15 (23) | 16 (21) | 18 (20) | 18 (21) | 33 (49)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 6 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 10 (12) | 9 (10) | 9 (9) | 10 (19) | 10 (10) | 5 (6)
Eructation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 5 (5) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 6 (6) | 0 (0) | 0 (0) | 12 (13)
Nausea (Gastrointestinal disorders) | 29 (40) | 35 (47) | 34 (40) | 39 (61) | 47 (76) | 8 (9)
Steatorrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (5)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 7 (9) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 6 (7) | 12 (15) | 13 (24) | 16 (20) | 13 (16) | 0 (0)
Fatigue (General disorders) | 8 (9) | 7 (7) | 8 (8) | 8 (8) | 13 (13) | 0 (0)
Oedema peripheral (General disorders) | 6 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 7 (7) | 5 (6) | 0 (0) | 6 (6)
Cystitis (Infections and infestations) | 6 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 13 (13) | 13 (16) | 20 (31) | 15 (19) | 21 (26) | 20 (24)
Gastroenteritis viral (Infections and infestations) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 10 (16) | 24 (37) | 11 (17) | 17 (23) | 22 (39) | 25 (39)
Nasopharyngitis (Infections and infestations) | 41 (85) | 37 (69) | 34 (71) | 42 (80) | 38 (74) | 26 (46)
Pharyngitis (Infections and infestations) | 5 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 8 (13) | 8 (10) | 8 (11) | 5 (10) | 6 (7)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (6)
Upper Respiratory Tract Infection (Infections and infestations) | 9 (13) | 10 (11) | 8 (16) | 12 (13) | 13 (20) | 13 (16)
Urinary Tract Infection (Infections and infestations) | 5 (8) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (6)
Joint sprain (Injury, poisoning and procedural complications) | 5 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 7 (8)
Blood insulin increased (Investigations) | 0 (0) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood TSH increased (Investigations) | 0 (0) | 0 (0) | 5 (7) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 14 (15) | 9 (10) | 0 (0) | 10 (12) | 5 (5) | 7 (9)
Back pain (Musculoskeletal and connective tissue disorders) | 14 (15) | 9 (10) | 16 (20) | 16 (17) | 12 (18) | 16 (21)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (5)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 5 (9) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 6 (6) | 0 (0) | 0 (0) | 7 (9) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 9 (10) | 5 (7) | 9 (9) | 6 (6) | 7 (8) | 6 (6)
Dizziness (Nervous system disorders) | 12 (12) | 7 (8) | 6 (8) | 6 (8) | 9 (9) | 0 (0)
Headache (Nervous system disorders) | 23 (37) | 23 (41) | 16 (23) | 23 (54) | 22 (25) | 16 (26)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 7 (8) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 7 (8) | 0 (0) | 0 (0) | 0 (0) | 6 (6)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 5 (5) | 0 (0) | 0 (0) | 7 (7) | 9 (10)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 7 (7) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Novo Nordisk acknowledges the Investigator's right to publish the entire results of the trial. Any such scientific paper, presentation, communication or other information concerning the investigation described in this protocol, must be submitted in writing to Novo Nordisk's Trial Manager prior to submission for publication/presentation for comments. Comments will be given within four weeks from receipt of the manuscript.